CLINICAL TRIAL: NCT00931268
Title: Morphological and Functional Evaluation of Buttock Lipoatrophy Treatment With Stabilized Hyaluronic Acid of Non-animal Origin (Macrolane); a Baseline-controlled Single-centre Study.
Brief Title: Morphological and Functional Evaluation of Buttock Lipoatrophy Treatment With Macrolane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31GC0804; AFFSAPS: 2008-A01252-53
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2013-11

CONDITIONS: Atrophy
Keywords: Lipoatrophy; Buttock treatment
MeSH Terms: conditions — Atrophy; Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macrolane VRF 30 (Other): Open label, baseline-controlled, one treatment session with injection of Macrolane VRF30 to each buttock, not exceeding 400 ml per subject.
  Interventions: Device: Macrolane VRF 30

INTERVENTIONS:
Device: Macrolane VRF 30 — One administration

SUMMARY:
The study is being undertaken to establish the effectiveness and safety of Macrolane volume restoration factor 30 (VRF30) when used for treatment of HIV-infected subjects with buttocks lipoatrophy.

ELIGIBILITY:
Inclusion Criteria:

* Have buttocks lipoatrophy and is unable to remain seated for more than 30 minutes due to pain.
* Have undergone HIV treatment for more than 2 years.
* Have RNA copies less than 50/ml.
* Have CD4 more than 200 cell/mm3.

Exclusion Criteria:

* Active infections.
* Active skin disease, inflammation or related conditions.
* Perineal pathology.
* Condition that may affect pain assessment.
* Skin with underlying fibrous tissue.
* BMI less than 19.
* Insufficient tissue cover in the area to be treated.
* Concomitant anticoagulant therapy and therapy with inhibitors of platelet aggregation within 14 days prior to treatment, or a history of bleeding disorders.
* Permanent implant placed in the treatment area.
* Other injectable implant, liposuction or other surgical therapy in the treatment area.
* Presence or history of connective tissue diseases.
* Tumors or pre-malign tissue disorder near or on the area to be treated.
* Contraindications for MRI
* Previous hypersensitivity to hyaluronic acid, or to the local anesthetic or antibiotic used in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Affairs, Study Director — Galderma R&D
Locations (1):
- Henri Mondor Hospital, Créteil, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled (screened) and treated: 11 August 2009. Last subject completed study: 2 September 2011.
Period: Overall Study
Arm/Group | Macrolane VRF 30
Started | 10
Completed | 4
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Macrolane VRF 30
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  France | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From 6 Months to Baseline in Visual Analogue Scale (VAS) Pain After 15 Minutes of Sitting
Description: Pain at sitting was evaluated using a 100 mm VAS with the descriptors 0 = "no pain" to the left and 100 = "worst possible pain" to the right. Pain was assessed by the subject after sitting 15 minutes on a standardized chair. The VAS pain at 6 months was compared to baseline and the change was calculated.
Time Frame: 6 months after treatment compared to baseline
Population: All efficacy analyses were performed using the intention to treat (ITT) population. The ITT population at baseline and 6 months comprised all 10 treated subjects.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Macrolane VRF 30
Number analyzed (Participants) | 10
mm | -28.1 (22.2)

2. Secondary Outcome: Change From up to 18 Months to Baseline in Visual Analogue Scale (VAS) Pain After 15 Minutes of Sitting
Description: Pain at sitting was evaluated using a 100 mm VAS with the descriptors 0 = "no pain" to the left and 100 = "worst possible pain" to the right. Pain was assessed by the subject after sitting 15 minutes on a standardized chair. The change in VAS pain was assessed at the time points 1, 3, 9, 12 and 18 months compared to baseline.
Time Frame: Baseline and up to 18 months after treatment
Population: The VAS pain at 1, 3, 9, 12 and 18 months after treatment was compared to baseline. Of 10 treated subjects the ITT populations at each time point was: 9 (1 month), 8 (3 months), 7 (9 months), 5 (12 months) and 4 (18 months).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Macrolane VRF 30
Number analyzed (Participants) | 10
mm
  VAS pain; change from 1 month to baseline | -14.3 (15.3)
  VAS pain; change from 3 months to baseline | -40.3 (8.9)
  VAS pain; change from 9 months to baseline | -29.4 (22.3)
  VAS pain; change from 12 months to baseline | -22.4 (25.2)
  VAS pain; change from 18 months to baseline | -15.8 (12.7)

3. Secondary Outcome: Quality of Life Assessed by MOS-HIV (Medical Outcome Study-HIV) Questionnaire
Description: A physical health summary score and a mental health summary score was generated on a rating scale of 0 to 100 where higher scores indicate better health. The change in health summary scores were assessed at the time points 3, 6, 9, 12 and 18 months compared to baseline.
Time Frame: Baseline and at 6 months after treatment
Population: The physical and mental health summary scores at 6 months after treatment were compared to baseline. The ITT population comprised 8 of 10 treated subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Macrolane VRF 30
Number analyzed (Participants) | 8
units on a scale
  Physical health; change from 6 months to baseline | 9.0 (6.2)
  Mental health; change from 6 months to baseline | 5.1 (15.6)

4. Secondary Outcome: Number of Participants With Global Esthetic Improvement
Description: Number of participants maintaining an improvement compared to baseline using the Global Esthetic Improvement Scale (GEIS) consisting of 5 grades (worse/no change/improved/much improved/very much improved), where the three latter indicates improvement. GEIS was assessed at the time points 1, 3, 6, 9, 12 and 18 months compared to pre-treatment photos.
Time Frame: One month and up to 18 months after treatment
Population: The ITT population at 6 months comprised all 10 treated subjects.
Measure: Number; unit: participants
Arm/Group | Macrolane VRF 30
Number analyzed (Participants) | 10
participants
  Subject assessed improvement at 6 months | 10
  Physician assessed improvement at 6 months | 10

5. Secondary Outcome: Number of Participants With Gel Displacement Evaluated by Magnetic Resonance Imaging (MRI)
Description: MRI was performed at baseline and at 1, 6, 9, and 12 months to determine the implant volume, thickness, localization and the possible local displacement of the implant. At the 6, 9 and 12 month visits any displacement was evaluated with MRI by comparison to the 1-month position of the gel. The number of participants with gel displacement are shown below.
Time Frame: 12 months after treatment
Measure: Number; unit: participants
Arm/Group | Macrolane VRF 30
Number analyzed (Participants) | 6
participants
  Gel displacement right buttock | 0
  Gel displacement left buttock | 0

6. Secondary Outcome: Adverse Event Recording
Description: Adverse events (AEs) were collected by open questioning, investigator findings, spontaneous reports and by direct questioning in the Case Report Form (CRF).
Time Frame: Up to 18 months after treatment
Population: Reported AEs, Safety population
Measure: Number; unit: participants
Arm/Group | Macrolane VRF 30
Number analyzed (Participants) | 10
participants | 3

7. Secondary Outcome: Time Until it Became Impossible to Stay Sitting
Description: Evaluation of when (in minutes) it became impossible for the subject to stay in the sitting position on a standardized chair, at the time points 1, 3, 6, 9, 12 and 18 months compared to baseline. In this analysis "more than 60 minutes" was handled as 60 minutes.
Time Frame: Baseline and at 6 months after treatment
Population: The ITT population at 6 months comprised all 10 treated subjects.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Macrolane VRF 30
Number analyzed (Participants) | 10
minutes
  Mean value at baseline | 23.8 (4.1)
  Mean value at 6 months | 59.0 (3.2)

ADVERSE EVENTS:
Time Frame: From treatment up to 18 months.
Description: Adverse events (AEs) were collected by open questioning, investigator findings, spontaneous reports and by direct questioning in the Case Report Form (CRF).
Arm/Group | Macrolane VRF 30
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macrolane VRF 30 (N=10)
Implant site effusion (General disorders) | 2 (2)
Injection site inflammation (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less